CLINICAL TRIAL: NCT03200717
Title: A Prospective International Multicenter Phase II Study to Evaluate the Efficacy, Safety and Quality of Life of Pazopanib in Patients With Advanced and/or Metastatic Renal Cell Carcinoma After Previous Therapy With Checkpoint Inhibitor Treatment
Brief Title: Study of Efficacy, Safety, and Quality of Life of Pazopanib in Patients With Advanced and/or Metastatic Renal Cell Carcinoma After Prior Checkpoint Inhibitor Treatment
Acronym: IO-PAZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPZP034A2410; 2017-000708-10 (EudraCT Number)
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Advanced Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
Keywords: renal cell carcinoma; metastatic renal cell; pazopanib; checkpoint inhibitor therapy; RCC; hypernephroma; renal adenocarcinoma; kidney cancer; renal cancer; adult
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pazopanib- 2nd line treatment (Experimental): Participants received pazopanib as 2nd line treatment
  Interventions: Drug: Pazopanib
- Pazopanib- 3rd line treatment (Experimental): Participants received pazopanib as 3rd line treatment
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Participants received 800mg of pazopanib once daily orally. Pazopanib was supplied as aqueous film-coated tablets containing 200 mg or 400 mg.

SUMMARY:
The main purpose of this study was to assess the progression-free survival (PFS) based on local investigator assessment of pazopanib in participants with advanced and/or metastatic renal cell carcinoma (mRCC) following prior treatment with immune checkpoint inhibitors (ICI).

DETAILED DESCRIPTION:
This was a multi-center, open-label, single-arm Phase II study to determine the efficacy, tolerability, safety and quality of life of treatment with pazopanib in subjects with advanced and/or metastatic renal cell carcinoma (RCC) following prior treatment with immune checkpoint inhibitors (ICI).

Subjects could have received prior systemic therapy with an ICI (monotherapy or combination) as 1st or 2nd line RCC treatment. However, they must not have received pazopanib previously. In this study, pazopanib could be administered in the 2nd or 3rd line setting. The therapeutic line for individual subjects was assigned at the time of screening.

Subjects received 800 mg of pazopanib daily until disease progression, unacceptable toxicity, death, pregnancy, start of a new anti-neoplastic therapy, discontinuation at the discretion of the investigator or patient, lost to follow-up or end of study, whichever came first.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed locally recurrent or metastatic predominantly clear cell renal cell carcinoma.
* Measurable disease based on RECIST 1.1 criteria
* Prior systemic therapy with an immune checkpoint inhibitor (monotherapy or combination) as 1st or 2nd line RCC treatment. Note: patients with prior mTOR inhibitor or TKI treatment as monotherapy or in combination with immune checkpoint inhibitor were allowed; however, treatment with immune checkpoint inhibitor (monotherapy or in combination) must have been the last treatment prior to study entry.
* Last dose of immune checkpoint inhibitor therapy received 4 or more weeks before start of study treatment
* Karnofsky performance status ≥70%.
* Potassium, sodium, calcium and magnesium within normal limits of the central laboratory

Key Exclusion Criteria:

* Renal cell carcinoma without any clear (conventional) cell component
* History or evidence of central nervous system (CNS) metastases (patients with pretreated metastases were eligible under certain conditions)
* Prior treatment with pazopanib
* Prior treatment with bevacizumab that was not given in combination with immune checkpoint inhibitor therapy.
* Prior treatment with more than 2 lines of therapy (combination treatments were considered 1 line of therapy)
* Not recovered from toxicity from prior immune checkpoint inhibitor therapy. Recovery was defined as ≤ NCI-CTCAE Grade 1, except for liver function test levels which must be <Grade 1.
* Disease recurrence less than 6 months from the last dose of prior neoadjuvant or adjuvant therapy (including VEGF-R TKI)
* Patients receiving prohibited concomitant medications that could not be discontinued or replaced by safe alternative medication at least 5 half-lives of the concomitant medication or 7 days, whichever was longer, prior to the start of pazopanib treatment.
* Administration of any investigational drug within 4 weeks prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Roswell Park Cancer Institute, Buffalo, New York, United States
- Novartis Investigative Site, Caba, Buenos Aires, Argentina
- Austria (3):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Calgary, Alberta, Canada
- Chile (2):
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, Santiago
- Czechia (2):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
- France (3):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Valenciennes
- Germany (3):
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Budapest, Hungary
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Madrid
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Preston

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 22 centers in 11 countries
Pre-assignment Details: A total of 87 participants were screened of which 62 participants were enrolled in the this study to receive study treatment.
Groups:
- Pazopanib- 2nd Line: Participants received pazopanib as 2nd line treatment
- Pazopanib- 3rd Line: Participants received pazopanib as 3rd line treatment
Period: Overall Study
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line
Started | 47 | 15
Completed | 6 | 0
Not Completed | 41 | 15
Not completed — Progressive disease | 24 | 5
Not completed — Adverse Event | 11 | 8
Not completed — Physician Decision | 3 | 2
Not completed — Death | 2 | 0
Not completed — Subject/Guardian Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | Total
Number analyzed (Participants) | 47 | 15 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (11.55) | 65.4 (9.77) | 63.2 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 36 | 11 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 13 | 57
  Asian | 1 | 0 | 1
  Other | 0 | 1 | 1
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the start date of pazopanib treatment to the date of the first documented progression or death due to any cause. PFS was assessed via local review according to RECIST 1.1.
  PFS was censored at the date of the last adequate tumor assessment if no PFS event (disease progression or death due to any cause) was observed prior to the analysis cut-off date.
  The PFS distribution was estimated using the Kaplan-Meier method.
Time Frame: Date of first treatment to date of progression or death up to approximately 38 months
Population: Full Analysis Set (FAS): all subjects to whom study treatment has been assigned and who received at least one dose of pazopanib.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Participants: All participants who received pazopanib as 2nd or 3rd line treatment
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | All Participants
Number analyzed (Participants) | 47 | 15 | 62
Months | 7.5 [3.7 to 12.6] | 4.6 [3.3 to 9.2] | 6.8 [3.7 to 11.1]

2. Secondary Outcome: Overall Response Rate (ORR) Based on Local Investigator Assessment According to RECIST v1.1
Description: ORR is defined as the percentage of participants with best overall response of confirmed complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST v1.1. The 95% confidence intervals (CIs) were computed using Clopper and Pearson method.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 38 months
Population: Full Analysis Set (FAS): All participants to whom study treatment was assigned and who received at least one dose of pazopanib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | All Participants
Number analyzed (Participants) | 47 | 15 | 62
Percentage of participants | 23.4 [12.3 to 38.0] | 0 [0.0 to 21.8] | 17.7 [9.2 to 29.5]

3. Secondary Outcome: Clinical Benefit Rate (CBR) Based on Local Investigator Assessment According to RECIST v1.1.
Description: CBR is defined as the percentage of participants with a best overall response of CR or PR or an overall lesion response of stable disease (SD) or Non-CR/Non-PD lasting ≥ 24 weeks based on local investigator's assessment according to RECIST v1.1. The 95% confidence intervals (CIs) were computed using Clopper and Pearson method.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 38 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | All Participants
Number analyzed (Participants) | 47 | 15 | 62
Percentage of participants | 53.2 [38.1 to 67.9] | 40.0 [16.3 to 67.7] | 50.0 [37.0 to 63.0]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first administration of study treatment until death due to any cause. If a participant was not known to have died, survival was censored at the date of last known date patient alive.
  The OS distribution was estimated using the Kaplan-Meier method.
Time Frame: From date of first treatment to date of death, up to approximately 44 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | All Participants
Number analyzed (Participants) | 47 | 15 | 62
Months | 27.8 [14.9 to NA] — NA: Not estimable due to insufficient follow-up time | 20.0 [9.2 to 25.6] | 23.4 [14.9 to 31.8]

5. Secondary Outcome: Duration of Response (DOR) Based on Local Investigators Assessment According to RECIST v1.1
Description: DOR is defined as the time from the date of first documented response (confirmed CR or PR according to RECIST v1.1 based on local Investigators review of tumor assessment data) to the date of tumor progression, or death due to underlying cancer, whichever comes first.
  If a patient not had an event, duration was censored at the date of last adequate tumor assessment.
  The DOR distribution was calculated using the Kaplan-Meier method.
Time Frame: From the date of first documented response (confirmed CR or PR) to the date of tumor progression, up to approximately 36 months
Population: Participants in the Full Analysis Set (FAS) for whom best overall response is complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line
Number analyzed (Participants) | 11 | 0
Months | NA [9.5 to NA] — NA: Not estimable due to insufficient number of participants with events |

6. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy- Kidney Symptom (FKSI-DRS) Score
Description: FKSI-DRS is a 9-item questionnaire specifically designed to evaluate symptoms that are directly attributable to kidney cancer and includes patient's symptoms in the past seven days such as lack of energy, pain, bone-pain, shortness of breath, fatigue, blood in urine, etc. Each item is scored on a 5-point scale (0=not at all to 4=very much). FKSI-DRS total score ranged from 0 (no symptoms) to 36 (most severe symptoms) with a higher score indicating greater presence of kidney cancer symptoms.
  The baseline is defined as the last FKSI-DRS assessment on or prior to first day of treatment.
  A negative change from baseline indicates improvement in kidney cancer symptom status.
Time Frame: Baseline, Day 1 of Cycle 2, 3, 4, 5, 6, 7, 9, 11, 13, 16 and every 3rd cycle thereafter until end of treatment, and end of treatment, assessed up to approximately 38 months. Cycle=28 days
Population: Full Analysis Set (FAS): All participants to whom study treatment was assigned and who received at least one dose of pazopanib. Number analyzed indicates participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | All Participants
Number analyzed (Participants) | 47 | 15 | 62
Score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 38 | 12 | 50
  Cycle 2 Day 1 | -1.3 (4.95) | -0.3 (4.31) | -1.0 (4.78)
  Cycle 3 Day 1: number analyzed (Participants) | 32 | 9 | 41
  Cycle 3 Day 1 | -0.5 (4.55) | 1.7 (4.18) | -0.0 (4.51)
  Cycle 4 Day 1: number analyzed (Participants) | 28 | 6 | 34
  Cycle 4 Day 1 | -0.1 (2.97) | 1.8 (4.22) | 0.2 (3.24)
  Cycle 5 Day 1: number analyzed (Participants) | 26 | 5 | 31
  Cycle 5 Day 1 | 0.1 (3.13) | 2.0 (2.35) | 0.4 (3.06)
  Cycle 6 Day 1: number analyzed (Participants) | 23 | 6 | 29
  Cycle 6 Day 1 | -0.3 (5.68) | 2.7 (3.27) | 0.3 (5.36)
  Cycle 7 Day 1: number analyzed (Participants) | 21 | 6 | 27
  Cycle 7 Day 1 | -0.1 (3.47) | 2.5 (3.73) | 0.4 (3.63)
  Cycle 9 Day 1: number analyzed (Participants) | 19 | 0 | 19
  Cycle 9 Day 1 | -0.1 (4.22) |  | -0.1 (4.22)
  Cycle 11 Day 1: number analyzed (Participants) | 16 | 1 | 7
  Cycle 11 Day 1 | 0.7 (3.30) | 0.0 (NA) — NA: The standard deviation was not estimable as there was only one participant. | 0.6 (3.20)
  Cycle 13 Day 1: number analyzed (Participants) | 10 | 0 | 10
  Cycle 13 Day 1 | 1.4 (2.12) |  | 1.4 (2.12)
  Cycle 16 Day 1: number analyzed (Participants) | 9 | 0 | 9
  Cycle 16 Day 1 | 0.6 (1.59) |  | 0.6 (1.59)
  Cycle 19 Day 1: number analyzed (Participants) | 6 | 0 | 6
  Cycle 19 Day 1 | 0.0 (2.76) |  | 0.0 (2.76)
  Cycle 22 Day 1: number analyzed (Participants) | 6 | 0 | 6
  Cycle 22 Day 1 | -0.5 (3.27) |  | -0.5 (3.27)
  Cycle 25 Day 1: number analyzed (Participants) | 4 | 0 | 4
  Cycle 25 Day 1 | 2.0 (2.31) |  | 2.0 (2.31)
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Cycle 31 Day 1: number analyzed (Participants) | 2 | 0 | 2
  Cycle 31 Day 1 | 0.5 (0.71) |  | 0.5 (0.71)
  Cycle 34 Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 34 Day 1 | 1.0 (NA) — NA: The standard deviation was not estimable as there was only one participant |  | 1.0 (NA) — NA: The standard deviation was not estimable as there was only one participant
  Cycle 37 Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 37 Day 1 | 1.0 (NA) — NA: The standard deviation was not estimable as there was only one participant |  | 1 (NA) — NA: The standard deviation was not estimable as there was only one participant
  End of Treatment: number analyzed (Participants) | 29 | 9 | 38
  End of Treatment | -0.6 (3.86) | -0.8 (6.00) | -0.6 (4.37)

7. Secondary Outcome: Change From Baseline in EuroQoL 5-level Instrument Visual Analogue Scale (EQ-5L-5D VAS) Score
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). The EQ-5L-5D VAS records the respondent's self-rated health on a vertical VAS, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state), with higher scores indicating higher health-related quality of life.
  The baseline is defined as the last EQ-5L-5D assessment on or prior to first day of treatment.
  A positive change from baseline indicates improvement in the heath state.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | All Participants
Number analyzed (Participants) | 47 | 15 | 62
Score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 38 | 12 | 50
  Cycle 2 Day 1 | 0.1 (16.44) | -1.9 (19.46) | -0.4 (17.02)
  Cycle 3 Day 1: number analyzed (Participants) | 30 | 9 | 39
  Cycle 3 Day 1 | -2.8 (14.35) | 3.6 (19.28) | -1.3 (15.58)
  Cycle 4 Day 1: number analyzed (Participants) | 28 | 6 | 34
  Cycle 4 Day 1 | -0.7 (10.88) | -1.5 (22.86) | -0.8 (13.27)
  Cycle 5 Day 1: number analyzed (Participants) | 25 | 5 | 30
  Cycle 5 Day 1 | -1.5 (13.61) | 3.2 (19.51) | -0.7 (14.45)
  Cycle 6 Day 1: number analyzed (Participants) | 23 | 6 | 29
  Cycle 6 Day 1 | -1.3 (18.35) | -3.5 (24.09) | -1.7 (19.21)
  Cycle 7 Day 1: number analyzed (Participants) | 21 | 6 | 27
  Cycle 7 Day 1 | 0.2 (11.89) | 0.7 (20.37) | 0.3 (13.73)
  Cycle 9 Day 1: number analyzed (Participants) | 19 | 0 | 19
  Cycle 9 Day 1 | 3.8 (11.64) |  | 3.8 (11.64)
  Cycle 11 Day 1: number analyzed (Participants) | 16 | 1 | 17
  Cycle 11 Day 1 | 3.9 (12.62) | -2.0 (NA) — NA: The standard deviation was not estimable as there was only one participant. | 3.5 (12.30)
  Cycle 13 Day 1: number analyzed (Participants) | 10 | 0 | 10
  Cycle 13 Day 1 | 5.7 (12.26) |  | 5.7 (12.26)
  Cycle 16 Day 1: number analyzed (Participants) | 9 | 0 | 9
  Cycle 16 Day 1 | -1.3 (11.70) |  | -1.3 (11.70)
  Cycle 19 Day 1: number analyzed (Participants) | 6 | 0 | 6
  Cycle 19 Day 1 | 5.5 (10.09) |  | 5.5 (10.09)
  Cycle 22 Day 1: number analyzed (Participants) | 6 | 0 | 6
  Cycle 22 Day 1 | 0.5 (9.93) |  | 0.5 (9.93)
  Cycle 25 Day 1: number analyzed (Participants) | 4 | 0 | 4
  Cycle 25 Day 1 | 0.0 (9.70) |  | 0.0 (9.70)
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Cycle 31 Day 1: number analyzed (Participants) | 2 | 0 | 2
  Cycle 31 Day 1 | 99.5 (0.71) |  | 99.5 (0.71)
  Cycle 34 Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 34 Day 1 | 10.0 (NA) — NA: The standard deviation was not estimable as there was only one participant. |  | 10.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  Cycle 37 Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 37 Day 1 | 90.0 (NA) — NA: The standard deviation was not estimable as there was only one participant. |  | 90.0 (NA) — NA: The standard deviation was not estimable as there was only one participant.
  End of Treatment: number analyzed (Participants) | 28 | 9 | 37
  End of Treatment | -1.9 (20.84) | -8.9 (19.99) | -3.6 (20.59)

8. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from first dose of study medication to 30 days after the last dose of study medication, for a maximum duration of approximately 38 months.
  Post-treatment survival follow-up deaths were collected from day 31 after last dose of study medication to end of study, up to approximately 44 months.
  All deaths refer to the sum of on-treatment deaths and post-treatment survival follow-up deaths.
Time Frame: On-treatment deaths: Up to approximately 38 months. Post-treatment survival follow-up deaths: Up to approximately 44 months
Population: Participants who received at least one dose of pazopanib
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib- 2nd Line | Pazopanib- 3rd Line | All Participants
Number analyzed (Participants) | 47 | 15 | 62
Participants
  On-treatment deaths | 5 | 1 | 6
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 35 | 13 | 48
  Post-treatment survival follow-up deaths | 22 | 10 | 32
  All deaths | 27 | 11 | 38

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days, up to a maximum duration of approximately 38 months. Deaths were collected in the post treatment survival follow up period from 31 days after last dose of study medication until the end of the study, up to approximately 44 months. These are not considered Adverse Events
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up.
  Deaths in the post treatment survival follow-up period are not considered Adverse Events. The total number at risk in the post treatment survival follow-up period includes patients that entered the post treatment survival follow-up period.
Groups:
- Pazopanib- 2nd Line (On-Treatment): AEs during on-treatment period (up to 30 days post-treatment)
- Pazopanib- 3rd Line (On-Treatment): AEs collected during on-treatment period (up to 30 days post- treatment)
- Pazopanib- 2nd Line (Post-treatment Survival Follow-up); Pazopanib- 3rd Line (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Pazopanib- 2nd Line (On-Treatment) | Pazopanib- 3rd Line (On-Treatment) | Pazopanib- 2nd Line (Post-treatment Survival Follow-up) | Pazopanib- 3rd Line (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 5/47 | 1/15 | 22/35 | 10/13
Serious Adverse Events (participants affected / at risk) | 21/47 | 9/15 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 46/47 | 14/15 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib- 2nd Line (On-Treatment) (N=47) | Pazopanib- 3rd Line (On-Treatment) (N=15) | Pazopanib- 2nd Line (Post-treatment Survival Follow-up) (N=0) | Pazopanib- 3rd Line (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Atrial flutter (Cardiac disorders) | 1 | 0 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 1 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 1 | NA | NA
Chest pain (General disorders) | 1 | 0 | NA | NA
Pyrexia (General disorders) | 2 | 0 | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 3 | 0 | NA | NA
Immune system disorder (Immune system disorders) | 0 | 1 | NA | NA
Bronchitis viral (Infections and infestations) | 0 | 1 | NA | NA
Meningitis bacterial (Infections and infestations) | 1 | 0 | NA | NA
Pulmonary sepsis (Infections and infestations) | 1 | 0 | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 1 | NA | NA
Viral infection (Infections and infestations) | 1 | 0 | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Alanine aminotransferase increased (Investigations) | 2 | 3 | NA | NA
Blood bilirubin increased (Investigations) | 1 | 0 | NA | NA
Transaminases increased (Investigations) | 1 | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | NA | NA
Dizziness (Nervous system disorders) | 1 | 0 | NA | NA
Spinal cord compression (Nervous system disorders) | 1 | 0 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 0 | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Hypertension (Vascular disorders) | 0 | 1 | NA | NA
Vasculitis (Vascular disorders) | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib- 2nd Line (On-Treatment) (N=47) | Pazopanib- 3rd Line (On-Treatment) (N=15) | Pazopanib- 2nd Line (Post-treatment Survival Follow-up) (N=0) | Pazopanib- 3rd Line (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | NA | NA
Hypothyroidism (Endocrine disorders) | 3 | 3 | NA | NA
Lacrimation increased (Eye disorders) | 0 | 1 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | NA | NA
Constipation (Gastrointestinal disorders) | 5 | 2 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 24 | 6 | NA | NA
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastritis (Gastrointestinal disorders) | 1 | 1 | NA | NA
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 12 | 4 | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | NA | NA
Stomatitis (Gastrointestinal disorders) | 6 | 2 | NA | NA
Vomiting (Gastrointestinal disorders) | 6 | 3 | NA | NA
Asthenia (General disorders) | 6 | 0 | NA | NA
Fatigue (General disorders) | 15 | 8 | NA | NA
Gait disturbance (General disorders) | 0 | 1 | NA | NA
Oedema peripheral (General disorders) | 3 | 1 | NA | NA
Pain (General disorders) | 0 | 1 | NA | NA
Peripheral swelling (General disorders) | 1 | 1 | NA | NA
Pyrexia (General disorders) | 3 | 1 | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 4 | 0 | NA | NA
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | NA | NA
Nasopharyngitis (Infections and infestations) | 2 | 1 | NA | NA
Rhinitis (Infections and infestations) | 0 | 1 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Alanine aminotransferase increased (Investigations) | 7 | 5 | NA | NA
Aspartate aminotransferase increased (Investigations) | 5 | 4 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | NA | NA
Blood bilirubin increased (Investigations) | 3 | 4 | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | NA | NA
Blood creatinine increased (Investigations) | 3 | 1 | NA | NA
Blood glucose increased (Investigations) | 0 | 1 | NA | NA
Blood urea increased (Investigations) | 0 | 1 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 3 | NA | NA
Lipase increased (Investigations) | 3 | 0 | NA | NA
Platelet count decreased (Investigations) | 0 | 1 | NA | NA
Serum ferritin increased (Investigations) | 0 | 1 | NA | NA
Transaminases increased (Investigations) | 2 | 1 | NA | NA
Troponin T increased (Investigations) | 0 | 1 | NA | NA
Weight decreased (Investigations) | 8 | 2 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 14 | 3 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | NA | NA
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA
Dizziness (Nervous system disorders) | 1 | 1 | NA | NA
Dysgeusia (Nervous system disorders) | 5 | 5 | NA | NA
Headache (Nervous system disorders) | 1 | 2 | NA | NA
Lethargy (Nervous system disorders) | 0 | 1 | NA | NA
Depression (Psychiatric disorders) | 1 | 1 | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 1 | NA | NA
Proteinuria (Renal and urinary disorders) | 3 | 2 | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 3 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | NA | NA
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Hypertension (Vascular disorders) | 13 | 3 | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT03200717/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03200717/SAP_001.pdf